CLINICAL TRIAL: NCT00553878
Title: Multi Center Double Blind Study Comparing 0.5 mg Dutasteride vs Placebo Daily in Men Receiving Intermittent Androgen Ablation Therapy for Prostate Cancer
Brief Title: Comparing 0.5 mg Dutasteride vs Placebo Daily in Men Receiving Androgen Ablation Therapy for Prostate Cancer
Acronym: AVIAS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Canadian Urology Research Consortium (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CURC/CUOG-AVIAS-0601; NCT00516815 (obsolete NCT alias)
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2012-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dutasteride (Placebo Comparator)
  Interventions: Drug: Dutasteride

INTERVENTIONS:
Drug: Dutasteride — dutasteride 0.5mg capsule daily until serum PSA rises to 5ng/ml in the off treatment interval
  Other Names: placebo

SUMMARY:
Patient on an intermittent androgen deprivation protocol for biochemical recurrence after radical local therapy for prostate cancer,the addition of continuous dutasteride treatment, significantly prolongs the duration of the off treatment interval and time to androgen independence.

DETAILED DESCRIPTION:
The study is to assess the effect of therapy with repeat oral daily dosing of dutasteride 05 mg on the length of the off treatment interval in men receiving intermittent androgen therapy for localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Age_>45and<_80
* Histological confirmed adenocarcinoma of prostate
* Has received external beam radiation,brachytherapy or radical prostatectomy for the treatment of prostate ca
* Candidate for intermittent androgen ablation
* Minimum of 3 PSA values above nadir taken at least 1 month apart
* Serum testosterone >_250ng/dl,ECOG 0 or 1
* Negative bone scan within 12 months of visit 1
* Able to swallow and retain oral medication

Exclusion Criteria:

* Previous treatment with chemotherapy
* Hormonal therapy with in last year
* Glucocorticoid with in last 3 months
* LHRH analogues with in previous year
* Ketoconazole
* Non Steroidal anti-androgens with in previous year
* Concurrent or previous use of Finasteride Dutasteride 5a reductase inhibitor anabolic steroids
* Over the counter or herbal prep such as saw palmetto selenium or vitamin E within last year
* May not be receiving any other investigational drug with in last 30 days
* Evidence of distant metastases
* Has received adjuvant or neoadjuvant ablation in past 12 months
* Unstable serious co-existing medical condition
* Abnormal liver and kidney functions
* Previous malignancy not including curative treated basal cell carcinoma of skin with in 5 years and bladder cancer with in past 2 years
* Known hypersensitivity to any 5a-reductase inhibitor or to any drug chemically related to dutasteride
* Known hypersensitivity to bicalutamide.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To assess whether repeat oral once daily dosing of dutasteride 0.5mg increases the length of the off treatment interval in men receiving intermittent androgen ablation therapy for localized prostate cancer | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Klotz, MD, Principal Investigator — CURC; Larry S Goldeng, Principal Investigator — CUOG
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
plan to share in publication